CLINICAL TRIAL: NCT02405416
Title: A Prospective Randomized Controlled Trial to Compare Infrahepatic Inferior Vena Cava Clamping With Selective Hepatic Vascular Exclusion Involving the Portal Triad Clamping in Hepatectomy
Brief Title: Infrahepatic Inferior Vena Cava Clamping Versus Selective Hepatic Vascular Exclusion Involving the Portal Triad Clamping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Chairman and Professor of Department of Surgery, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: chenxp006; 2012ZX10002016-004 (Other Grant/Funding Number: The State Key Project on Inflection Disease of China)
Record Dates: First submitted 2015-03-07; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Liver Neoplasms; Liver Cirrhosis
Keywords: Hepatocellular Carcinoma; Blood Loss; Haemorrhage; Vascular Control
MeSH Terms: conditions — Liver Neoplasms; Liver Cirrhosis; Carcinoma, Hepatocellular; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IIVCC group (Experimental): The portal triad and infrahepatic inferior vena cava are dissected and taped with a vessel loop, respectively. During liver parenchymal resection，portal triad and infrahepatic inferior vena cava clampings are performed at the specified transection depth from liver surface successively.
  Interventions: Procedure: Infrahepatic inferior vena cava clamping; Procedure: Portal triad clamping
- SHVE group (Active Comparator): In this group, the portal triad clamping and selective hepatic vascular exclusion of major hepatic veins are used. Different major hepatic veins are occluded by clamping forcep depending on the site of tumors. The clamping timepoints are same as the IIVCC group.
  Interventions: Procedure: Selective hepatic vascular exclusion; Procedure: Portal triad clamping

INTERVENTIONS:
Procedure: Infrahepatic inferior vena cava clamping — Infrahepatic inferior vena cava is clamped in hepatectomy.
  Other Names: IIVCC
  Arms: IIVCC group
Procedure: Selective hepatic vascular exclusion — Selected major hepatic vein is clamped in hepatectomy.
  Other Names: SHVE
  Arms: SHVE group
Procedure: Portal triad clamping — Portal triad are clamped in hepatectomy.
  Other Names: PTC

SUMMARY:
This clinical trial aims to compare infrahepatic inferior vena cava clamping (IIVCC) with selective hepatic vascular exclusion (SHVE) involving the portal triad clamping (PTC) in complex cirrhotic liver resection. One group will receive IIVCC plus PTC, while an another equivalent group patients will be operated using SHVE and PTC.

DETAILED DESCRIPTION:
Intraoperative blood loss is significantly associated with clinical outcomes of patients undergoing hepatectomy. There have been various hepatic vascular control techniques, including infrahepatic inferior vena cava clamping (IIVCC) and selective hepatic vascular exclusion (SHVE).The propose of this study is to compare these two surgical techniques combined with the portal triad clamping (PTC) in hepatic cirrhotic patients. All patients being performed hepatectomy at the center are scanned according to inclusion and exclusion criteria. After intraoperative exploration, patients are randomized into two interventional groups. PTC, IIVCC or SHVE is performed at the specified timepoint in liver parenchymal transection in two different groups. All data are collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. either male or female, older than 18 (include 18).
2. tumors oppress or be in close proximity to one or more of major hepatic veins.
3. the maximum diameter of tumor ≥ 5cm, number of lesions ≤ 3 and should be in same liver lobe if multiple lesions exit.
4. preoperative liver function assessment: Child-Pugh classification is A or B.
5. preoperative laboratory test: blood platlet count > 100×10^9/l, prothrombin activity > 60%.
6. liver cirrhosis.

Exclusion Criteria:

1. contraindication for surgery,e.g.severe disorders of circulation, respiratory or renal system.
2. extrahepatic metastasis in patients with malignancy or tumor invasion of portal vein, hepatic vein, bile duct or inferior vena cava.
3. hepatectomy accompanied with other organs resection(e.g. bile duct, intestine, pancreas or stomach)
4. regular hepatectomy.
5. tumors located in the left lateral lobe of liver.
6. previous hepatectomy.
7. pregnancy or lactation.
8. refusal to participate this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | Intraoperative period
  blood loss from incision to closure
Normalized transection-related blood loss | Intraoperative period
  Intraoperative blood loss normalized by transection surface area

SECONDARY OUTCOMES:
Time of infrahepatic inferior vena cava or selected hepatic vein dissection | Intraoperative period
  Time cost of dissection
Variations of intraoperative infrahepatic inferior vena cava pressure or hepatic vein pressure | Intraoperative period
Drop of hemoglobin level | Drop of hemoglobin level will be measured during liver parenchymal transection period(neither the specific time point nor expected average could be given prospectively because of different surgical situations)
Postrecovery of liver function | postoperative days 1, 3, 5, 7
  Liver function evaluation is composite of liver enzyme ，total bilirubin, prothrombin activity, etc.
Postrecovery of renal function | postoperative days 1, 3, 5, 7
  Renal function evaluation is composite of blood urea nitrogen, creatinine, etc.
Morbidity of postoperative complications | 90 days after surgery
Postoperative mortality | 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, M.D., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China